CLINICAL TRIAL: NCT06794073
Title: Efficacy and Safety of Multimodal Ablation Combined With PD-1 Monoclonal Antibody, Lenvatinib and TACE in the Treatment of Unresectable Primary Hepatocellular Carcinoma: A Single-Arm, Single-Center Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTT-B2024
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Hepatocellular; Neoplasms, Glandular and Epithelial; Adenocarcinoma; Digestive System Neoplasms; Liver Neoplasms
Keywords: Multimodal; Tislelizumab; lenvatinib; TACE; unresectable primary liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms, Glandular and Epithelial; Adenocarcinoma; Digestive System Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): The patient will receive induction therapy with tislelizumab and lenvatinib within 14 days after enrollment. Subsequently, within 2-7 days (the exact timing will be determined based on clinical circumstances), they will undergo Multimodal Thermal Therapy (MTT). Following the MTT procedure, on-demand TACE treatment will be administered. Starting from day 7 post-MTT (with the exact timing adjusted according to clinical conditions), the patient will resume tislelizumab and lenvatinib therapy until disease progression, occurrence of intolerable toxicity, or withdrawal of consent.
  Interventions: Device: Multimodal Thermal Therapy

INTERVENTIONS:
Device: Multimodal Thermal Therapy — The high-burden tumor is identified as the target lesion for treatment. A pre-treatment biopsy of the target lesion is performed to obtain tumor tissue. Multimodal ablation therapy of the target lesion is conducted under CT guidance. The treatment procedure follows the tumor ablation protocol using the multimodal therapy radiofrequency temperature-controlled mode.

SUMMARY:
This study is a prospective, single-arm, single-center trial evaluating the efficacy of TACE combined with multimodal ablation, Tislelizumab, and lenvatinib in the treatment of unresectable primary liver cancer.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of multimodal ablation combined with Tislelizumab, lenvatinib, and TACE in the treatment of primary liver cancer. By comparing preoperative and postoperative immune markers, the study seeks to clarify the clinical value of multimodal ablation combined with systemic therapy and TACE in the management of primary liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, regardless of gender.
2. Clinically or pathologically confirmed HCC.
3. CNLC stage IIb-IIIa, deemed unresectable after multidisciplinary evaluation.
4. No prior systemic chemotherapy, targeted therapy, or immunotherapy for HCC, or prior-treated patients with a best response of SD or PD.
5. At least one measurable, untreated lesion eligible for ablation, with the largest target lesion diameter >5 cm.
6. ECOG PS 0-1 and an expected survival >3 months.
7. Child-Pugh score ≤7.

Exclusion Criteria:

1. Child-Pugh class C liver dysfunction.
2. Tumor thrombus in the main portal vein or hepatic vein.
3. Extensive metastatic disease with an expected survival <3 months.
4. Severe dysfunction of major organs (liver, kidney, heart, lung, or brain).
5. History of esophageal/gastric variceal bleeding within the past month.
6. History of other malignancies.
7. Last anti-tumor therapy (e.g., radiotherapy, systemic chemotherapy, or local treatment) within <1 month.
8. Active infection; HBV co-infection (HBV DNA ≥2000 IU/mL or ≥10⁴ copies/mL unless reduced by one log after antiviral therapy); HCV co-infection requiring guideline-directed antiviral treatment; HIV infection; or biliary tract inflammation.
9. History of organ transplantation or hepatic encephalopathy.
10. Uncorrectable coagulation disorders.
11. Refractory massive ascites, pleural effusion, or cachexia.
12. Pregnancy, impaired consciousness, or inability to comply with treatment.
13. High tumor burden (sum of the largest liver lesion diameter and number of liver lesions >12).
14. Any other condition deemed unsuitable by investigators that may affect study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to RECIST 1.1 and mRECIST | Follow-up for 12 months, with evaluations conducted at 2 weeks, 6 weeks, 3 months, 6 months, 9 months, and 12 months postoperatively.
  Refers to the proportion of patients whose tumors shrink to a certain extent and maintain that response for a specified period, including cases of Complete Response (CR) and Partial Response (PR). Tumor objective response is assessed using RECIST 1.1 and mRECIST criteria. At baseline, subjects must have measurable tumor lesions. According to the efficacy evaluation criteria, the outcomes are classified as Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD).

SECONDARY OUTCOMES:
Progression-Free Survival（PFS） | Follow-up for 12 months,with assessments conducted every 3 months.
  It refers to the time from the date of enrollment to the date of the first recorded disease progression(PD)or death,whichever occurs first.
Overall Survival（OS） | Follow-up for 12 months,with assessments conducted every 3 months.
  Overall Survival(OS)refers to the time from the date of enrollment to the date of death due to any cause.
Safety and Tolerability | Follow-up for 12 months, with evaluations conducted at 2 weeks, 6 weeks, 3 months, 6 months, 9 months, and 12 months postoperatively.
  Safety:Refers to the extent to which a drug does not cause unacceptable harm or side effects when applied in the human body.Tolerability:Refers to the degree to which patients accept the side effects that occur after treatment,reflecting their ability to endure the side effects of the medication.All adverse events will be recorded and assessed for severity based on the NCI-CTC AE 5.0 grading criteria.During the follow-up period,all subjects will be continuously monitored,and the occurrence,duration,severity,and treatment-relatedness of adverse events will be documented.

IPD SHARING:
Plan to Share IPD: No